CLINICAL TRIAL: NCT06347744
Title: Radicle Rest™ 24: A Randomized, Double-Blind, Placebo-Controlled Direct-to-Consumer Study Assessing the Impact of Health and Wellness Products on Sleep and Related Health Outcomes
Brief Title: Radicle Rest 24: A Study of Health and Wellness Products on Sleep and Related Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX-P-2401
Record Dates: First submitted 2024-03-28; First posted 2024-04-04 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-03

CONDITIONS: Sleep; Sleep Disturbance; Sleep Disorder
MeSH Terms: conditions — Parasomnias; Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be stratified based on gender at birth then randomized to one of the study arms.
Who Masked: Participant, Investigator
Masking Description: Participants will be stratified based on gender at birth then randomized to one of the study arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Placebo Control 1 (Placebo Comparator): Rest Product Form 1 - control
  Interventions: Dietary Supplement: Radicle Rest Placebo Control Form 1
- Active Product 1.1 (Experimental): Rest Product Form 1 - active product 1
  Interventions: Dietary Supplement: Radicle Rest Active Study Product 1.1 Usage
- Placebo Control 2 (Placebo Comparator): Rest Product Form 2 - control
  Interventions: Dietary Supplement: Radicle Rest Placebo Control Form 2
- Active Product 2.1 (Experimental): Rest Product Form 2 - active product 1
  Interventions: Dietary Supplement: Radicle Rest Active Study Product 2.1 Usage
- Placebo Control 4.1.0 (Experimental): Rest Product 4 - control
  Interventions: Dietary Supplement: Radicle Rest Placebo Control 4.1.0
- Active Product 4.1.1 (Experimental): Rest Product 4 - active product 1
  Interventions: Dietary Supplement: Radicle Rest Active Study Product 4.1.1 Usage

INTERVENTIONS:
Dietary Supplement: Radicle Rest Placebo Control Form 1 — Participants will use their Radicle Rest Placebo Control Form 1 as directed for a period of 6 weeks.
  Arms: Placebo Control 1
Dietary Supplement: Radicle Rest Active Study Product 1.1 Usage — Participants will use their Radicle Rest Active Study Product 1.1 as directed for a period of 6 weeks.
  Arms: Active Product 1.1
Dietary Supplement: Radicle Rest Placebo Control Form 2 — Participants will use their Radicle Rest Placebo Control Form 2 as directed for a period of 6 weeks.
  Arms: Placebo Control 2
Dietary Supplement: Radicle Rest Active Study Product 2.1 Usage — Participants will use their Radicle Rest Active Study Product 2.1 as directed for a period of 6 weeks.
  Arms: Active Product 2.1
Dietary Supplement: Radicle Rest Placebo Control 4.1.0 — Participants will use their Radicle Rest Active Study Product 4.1.1 as directed for a period of 6 weeks.
  Arms: Placebo Control 4.1.0
Dietary Supplement: Radicle Rest Active Study Product 4.1.1 Usage — Participants will use their Radicle Rest Active Study Product 4.1.1 as directed for a period of 6 weeks.
  Arms: Active Product 4.1.1

SUMMARY:
A randomized, double-blind, placebo-controlled study assessing the impact of health and wellness products on sleep and related health outcomes.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study conducted with adult participants, residing in the United States.

Eligible participants will (1) endorse a desire for better sleep, (2) have the opportunity for meaningful improvement (at least 20%) in their primary health outcome, and (3) express acceptance in taking a product and not knowing its formulation until the end of the study.

Participants that report a known cardiac dysfunction, liver or kidney disease may be excluded. Participants that report a known contraindication or with well-established, significant safety concerns due to illness will be excluded. Heavy drinkers and those who report they are pregnant, trying to become pregnant, or breastfeeding will be excluded. Participants that report taking medications with a known contraindication or with well-established, significant safety concerns will be excluded.

Self-reported data are collected electronically from eligible participants for 7 weeks. Participant reports of health indicators will be collected at baseline, throughout the active period of study product use, and in a final survey. All study assessments will be electronic; there are no in-person visits or assessments for this real-world evidence study.

ELIGIBILITY:
Inclusion Criteria:

* Adults, at least 21 years of age at the time of electronic consent, inclusive of all ethnicities, races, and gender identities. Assigned sex at birth will determine sex-specific recruitment and surveys (male vs female) employed, when needed
* Resides in the United States
* Endorses better sleep as a primary desire
* Has the opportunity for at least 20% improvement in their primary health outcome
* Expresses a willingness to take a study product and not know the product identity (active or placebo) until the end of the study

Exclusion Criteria:

* Report being pregnant, trying to become pregnant, or breastfeeding
* Unable to provide a valid US shipping address and mobile phone number
* Reports current enrollment in another clinical trial
* Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day)
* Unable to read and understand English
* Reports a current and/or recent (up to 3 months ago) major illness and/or surgery that poses a known, significant safety risk.
* Reports a diagnosis of cardiac dysfunction, liver or kidney disease that presents a known contraindication and/or a significant safety risk with any of the study product ingredients. NYHA (New York Heart Association) Class Ill or IV congestive heart failure, atrial fibrillation, uncontrolled arrhythmias, cirrhosis, end-stage liver disease, stage 3b or 4 chronic kidney disease, or kidney failure
* Reports taking medications that have a well-established moderate or severe interaction, posing a substantial safety risk with any of the study product ingredients. Anticoagulants, antihypertensive, anxiolytics, antidepressants, chemotherapy, immunotherapy, sedative hypnotics, seizure medications, medications that warn against grapefruit consumption, corticosteroids at doses greater than 5 mg per day, diabetic medications, oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection, antipsychotics, MAOls (monoamine oxidase inhibitors), or thyroid products
* Reports current use of the primary ingredient(s) and/or similar product(s) to the active study product(s) that may limit the effects of the study products
* Lack of reliable daily access to the internet

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1646 (Actual)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Change in sleep | 6 weeks
  Mean difference in sleep score as assessed by Patient Reported Outcome Measurement System (PROMIS) Sleep Disturbance Short Form 8A (scale 8-40; where higher scores correspond to greater sleep disturbance)

SECONDARY OUTCOMES:
Change in feelings of anxiety | 6 weeks
  Mean difference in anxiety score as assessed by Patient Reported Outcome Measurement System (PROMIS) Anxiety 4A (scale 4-20; with higher scores corresponding to more severe anxiety)
Change in fatigue | 6 weeks
  Mean difference in fatigue score as assessed by Patient Reported Outcome Measurement System (PROMIS) Fatigue 4A (scale 4-20; where higher scores correspond to more severe fatigue)
Change in mood (emotional distress-depression) | 6 weeks
  Mean difference in emotional distress score as assessed by Patient Reported Outcome Measurement System (PROMIS) Emotional Distress- Depression 4A (scale 4-20; with higher scores corresponding to greater levels of emotional distress)
Minimal clinically important difference (MCID) in sleep | 6 weeks
  Likelihood of experiencing minimal clinically important difference in sleep score as assessed by Patient Reported Outcome Measurement System (PROMIS) Sleep Disturbance Short Form 8A (scale 8-40; where higher scores correspond to greater sleep disturbance)
Minimal clinically important difference (MCID) in feelings of anxiety | 6 weeks
  Likelihood of experiencing minimal clinically important difference in feelings of anxiety score as assessed by Patient Reported Outcome Measurement System (PROMIS) Anxiety 4A (scale 4-20; with higher scores corresponding to more severe anxiety)
Minimal clinically important difference (MCID) in fatigue | 6 weeks
  Likelihood of experiencing minimal clinically important difference in fatigue score as assessed by Patient Reported Outcome Measurement System (PROMIS) Fatigue 4A (scale 4-20; where higher scores correspond to more severe fatigue)
Minimal clinically important difference (MCID) in mood (emotional distress-depression) | 6 weeks
  Likelihood of experiencing minimal clinically important difference in mood score as assessed by Patient Reported Outcome Measurement System (PROMIS) Emotional Distress- Depression 4A (scale 4-20; with higher scores corresponding to greater levels of emotional distress)

CONTACTS AND LOCATIONS:
Overall Officials: Emily K. Pauli, PharmD, Principal Investigator — Radicle Science Inc.
Locations (1):
- Radicle Science, Inc, Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Radicle Science, Inc — http://radiclescience.com